CLINICAL TRIAL: NCT03189303
Title: Planned vs. Actual Acetabular Cup Position in Total Hip Arthroplasty With Standard Instrumentation and Technique
Brief Title: Cup Position in THA With Standard Instruments
Status: Completed | Type: Observational
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: DSJ_15010
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post Traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Primary Uncemented Total Hip Arthroplasty — The study devices are the Pinnacle Hip System acetabular cup with a Summit, Actis, or Corail femoral stem

SUMMARY:
Prospective, global, multicenter study to assess cup position in THA. After written informed consent has been obtained, study evaluations will be collected from the pre-op clinic visit, the operative visit (including discharge), and 6 and 12 weeks postoperatively.

DETAILED DESCRIPTION:
This is a global, prospective, multi-center study with a planned analysis of a minimum of 176 Subjects. Up to 15 study sites will participate in this study. The primary and secondary endpoints are as follows:

Primary endpoint:

The primary endpoint is acetabular cup position success at 6 weeks postoperatively. Success is defined as cup inclination and version within 10 degrees of the plan.

Secondary endpoints:

1. Inclination success (as defined for the primary endpoint)
2. Version success (as defined for the primary endpoint)
3. 90-day complication rates
4. Change from preoperative baseline for the Harris Hip Score
5. Radiographic Outcomes (based upon: AP Hip, AP Pelvis, and Modified Lauenstein Lateral)
6. Change from preoperative baseline for the EQ-5D-5L (health state, EQ-VAS, and index value, if applicable)
7. Change from 6 week baseline for the Forgotten Joint Score

ELIGIBILITY:
Inclusion Criteria:

1. All devices are to be used according to the approved indications
2. The patient is undergoing a standard of care hip replacement with the Pinnacle cup and a Corail, Summit, or Actis stem via the posterolateral, anterolateral, or direct lateral approach with the patient in the lateral decubitus position.
3. Individuals who are able to speak, read, and comprehend the Informed Consent Document and willing and able to provide informed patient consent for participation in the study and have authorized the transfer of his/her information to DePuy Synthes.
4. Individuals who are willing and able to complete follow-up as specified by the study protocol.
5. Individuals who are willing and able to complete the Subject Hip Outcomes questionnaires (i.e., FJS-12, EQ-5D-5L and Hip Evaluation) as specified by the study protocol.
6. Individuals who are not bedridden.
7. Individuals who are a minimum age of 21 years at the time of consent.

Exclusion Criteria:

1. Active local or systemic infection.
2. Loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the procedure unjustified.
3. Poor bone quality, such as osteoporosis, where, in the surgeon's opinion, there could be considerable migration of the prosthesis or a significant chance of fracture of the femoral shaft and/or the lack of adequate bone to support the implant(s).
4. Charcot's or Paget's disease.
5. The Subject is a woman who is pregnant or lactating.
6. Subject had a contralateral amputation.
7. Previous partial hip replacement in affected hip.
8. Subject has participated in a clinical investigation with an investigational product (drug or device) in the last three months.
9. Contralateral hip was replaced less than 6 months prior to surgery date
10. Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
11. Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
12. Subject has a medical condition with less than 2 years of life expectancy.
13. Subject, in the opinion of the Investigator, is a drug or alcohol abuser or has a psychological disorder that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who the investigator deems to be a candidate for a primary total hip arthroplasty (THA) using the study devices (Pinnacle cup with a Corail or Summit stem) in a primary uncemented THA.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Composite success of cup inclination and cup version. | 6 weeks
  The primary endpoint is acetabular cup position success at 6 weeks postoperatively. It is a composite endpoint; in order for an individual cup position to be considered successful, the cup's placement must satisfy all of the following criteria at 6 weeks:
  1. Inclination Success: within 10 degrees of the planned inclination
  2. Version Success: within 10 degrees of the planned version

SECONDARY OUTCOMES:
Inclination success | 6 weeks
  Inclination Success: within 10 degrees of the planned inclination
Version success | 6 weeks
  Version success: within 10 degrees of the planned version
90 day postoperative complication rates | 90 days postoperative
  The number of subjects and the percentage of subjects with complications at 90 days post-operatively
Harris Hip Score | Baseline and 6 and 12 weeks postoperative
  Change from preoperative baseline for the Harris Hip Score
Forgotten Joint Score | 6 and 12 weeks postoperative
  Change from 6 week baseline for the Forgotten Joint Score
EQ-5D-5L dimension score | Baseline and 6 and 12 weeks postoperative
  Mean change from baseline for the specified time points
EQ-VAS score (subscore of EQ-5D-5L) | Baseline and 6 and 12 weeks postoperative
  Mean change from baseline for the specified time points
EQ-5D-5L index value (if applicable) | Baseline and 6 and 12 weeks postoperative
  Mean change from baseline for the specified time points
Radiographic Outcomes | Baseline and 6 and 12 weeks postoperative
  Radiographs will be read by an independent radiographic reviewer (IRR) at 6 weeks to act as a baseline measurement to be compared to radiographs taken at later time points (12 weeks). Parameters measured include subsidence, migration, inclination and version angles, osteolysis, and radiolucency.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Mount Sinai Hospital, New York, New York
  - Carolina Orthopaedic and Sports Medicine Center, Gastonia, North Carolina
  - Orthopedic Specialists and Sports Medicine, Newark, Ohio
  - Lowcountry Orthopaedics & Sports Medicine, Charleston, South Carolina
- Istituto Orthopedico Galeazzi IRCCS, Milan, Italy
- Netherlands (3):
  - Bravis Hospital, Bergen op Zoom
  - Maastricht University Medical Center, Maastricht
  - Canisius Wilhelmina Hospital, Nijmegen
- United Kingdom (2):
  - Woodend Hospital, Aberdeen, Scotland
  - Glan Clwyd Hospital, Rhyl, Wales

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fawley D, Bernard T, Thomason HC 3rd, Zagra L, Ten Broeke RHM, Johnson K. Early functional recovery outcomes and return to work after primary total hip arthroplasty: a novel patient reported outcomes questionnaire. J Orthop Surg Res. 2024 Jul 26;19(1):434. doi: 10.1186/s13018-024-04937-z. PMID 39061099
- [Derived] Meermans G, Fawley D, Zagra L, Ten Broeke RHM, Johnson K, Bernard T, Thomason HC 3rd. Accuracy of cup placement compared with preoperative surgeon targets in primary total hip arthroplasty using standard instrumentation and techniques: a global, multicenter study. J Orthop Traumatol. 2024 May 10;25(1):25. doi: 10.1186/s10195-024-00766-2. PMID 38727945